CLINICAL TRIAL: NCT02739048
Title: Changes of Immunologic Function in Patients of Prostate Cancer Induced After Cryoablation.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jian Kang, Chief Physician, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-16-011
Record Dates: First submitted 2016-04-12; First posted 2016-04-14 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
1. The overall objective of the study: By evaluating the curative effect of CSAP in localized prostate cancer, locally advanced prostate cancer and metastasis advanced prostate cancer, and the change of state in cellular immunity and humoral immunity before and after CSAP. Validate the clinical therapeutic effect of all kinds of prostate cancer, as well as the change of immune status before and after CSAP.

2. The main content of the study:

1. Included in the samples are patients in hospitals for CSAP. The sample capacity are planned to be 80. The main purpose of the study is to observe the overall survival rate , disease free survival rate, the progress time of the PSA biochemical recurrence as well as the disease progress time.
2. Measure the change of concentration in peripheral blood T lymphocyte subsets (CD3 + T, CD4 + T, CD8 + T, CD4 + / CD8 + T, NK cells) and regulatory T cells before and after cryoablation within 1 month, 3 months and 6 months.
3. Measure the change of concentration in peripheral blood IFN-1, IL-4, IFN-1/IL-4 ratio (Thl/Th2 ratio), and detect the secretion of CD4 + Th tumor-specific IFN-l and the activity of tumor-specific killer CD8 + CTL before and after cryoablation within 2 weeks and 1 month.
4. Before cryoablation, detect the expression and distribution of Follistatin-Like1 (FSTL-1), Besides, verify the connection between the number and activation ratio of tumor local dendritic cells (DC) and the FSTL-1, evaluating the cryoablation effect on the immune response.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with prostate cancer by pathology
* the age of patients should be from 40 to 80 years old
* do not receive other treatments like radical prostatectomy, radiotherapy, etc

Exclusion Criteria:

* can not receive surgery because of bad performance status
* abnormal coagulation function
* receive other treatment before CSAP
* do not want to achieve CSAP because of any reasons

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 patients diagnose with prostate
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
humoral immunity and cellular immunity will be activated after CSAP for patients of prostate cancer | 3 years
  All 80 participants' peripheral blood will be collected before CSAP and after CSAP to detect the concentration of T lymphocyte subsets (CD3 + T, CD4 + T, CD8 + T, CD4 + / CD8 + T, NK cells), IFN-1, IL-4, IFN-1/IL-4 ratio (Thl/Th2 ratio) and FSTL-1, and to comment the change of activity of humoral immunity and cellular immunity.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Kang, director, Study Director — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided